CLINICAL TRIAL: NCT01602016
Title: A Folinic Acid Intervention for ASD: Links to Folate Receptor-alpha Autoimmunity & Redox Metabolism
Brief Title: A Folinic Acid Intervention for Autism Spectrum Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Non-compliance
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136002
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Autism Spectrum Disorder; Autistic Disorder; Autism; Asperger's Syndrome; Pervasive Development Disorders
Keywords: ASD; PDD-NOS
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive | interventions — Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I (No Intervention): Baseline Visit Phase 1: The screening portion of the CELF will be administered to the child to screen for language impairment. If a child is determined to be pre-verbal they will automatically qualify,If there is no language impairment, the subject will not be eligible. If language impairment is confirmed, the participant will immediately go on to the baseline visit of Phase 2.
- Phase II: 12 week Folinic Acid or Placebo intervention (Other): The child will be consented for Phase 2 (the RCT) and undergo a blood draw (up to 20mL) for metabolic and autoantibody testing. the child will undergo language and behavioral assessment while the parent will be interviewed for the Vineland and other questionnaires (ASQ, RBS-R, SRS, and ABC). Demographic information including; age, race, gender, and ethnicity will be collected. The research pharmacist will randomize the participant to either Intervention A or B (only the research pharmacist will know which intervention has the folinic acid). The research pharmacist will distribute the drug or placebo to the parent and instruct the parent of the proper administration of the intervention. This will be considered the 12 week randomly controlled clinical trial that is investigating the safety and efficacy of folinic acis interventions in ASD and will last for approximately 12 weeks. At the end of 12 weeks, the same assessments that were conducted at baseline will be readministered
  Interventions: Drug: Folinic Acid and placebo
- Phase III: Open Label Extension of Folinic Acid (Experimental): If consent for Phase 3 is signed by parents with children who qualify for Phase 3, the research pharmacist will provide a 12 week supply of folinic acid to the parent. This arm will be offered to all clients that completed phase 2 of the trial. After consenting and 12 weeks of folinic acid dosing, the client will come back and complete the same protocol and be tested on the same measures used in phase II of the study. This will be a rolling stopping point so that new therapies can be started, if the parent/caregiver is so inclined
  Interventions: Drug: Folinic Acid

INTERVENTIONS:
Drug: Folinic Acid and placebo — Capsules of folinic acid and placebo will be administered in 1mg/kg/day in two divided doses (0.5mg/kg/dose; 25mg/day maximum) for two weeks followed by 2 mg/kg/day with a maximum dose of 50mg/day provided the lower dose is well tolerated for 10 weeks.
  Arms: Phase II: 12 week Folinic Acid or Placebo intervention
Drug: Folinic Acid — capsules of folinic acis will be provided. The target dose will be 1mg/kg/day in two divided doses (0.5mg/kg/dose; 25mg/day maximum) for two weeks followed by 2 mg/kg/day with a maximum dose of 50mg/day provided the lower dose is well tolerated, for 10 weeks.
  Arms: Phase III: Open Label Extension of Folinic Acid

SUMMARY:
Researchers at Arkansas Children's Hospital Research Institute are conducting a study looking at the effects of Folinic Acid on language in Autism Spectrum Disorder and language impairment. The study has 3 phases. Phase 1 confirms that your child has language impairment (there is no compensation for this visit). If language impairment is verified in the phase 1 screening, then your child will be eligible for phase 2. Phase 2 consists of receiving 12 weeks of folinic acid or an inactive placebo, in addition to several evaluations of your child's abilities and a single blood test. Children that complete phase 2 will be eligible for a 12 week open-label trial of folinic acid which is phase 3.

DETAILED DESCRIPTION:
Evidence-based interventions for autism spectrum disorders (ASD) are limited. Currently, there is no FDA approved medical therapy that addresses either core ASD symptoms or pathophysiological processes associated with ASD. For example, the two FDA approved antipsychotic medications for treating ASD are indicated for symptoms associated with ASD, not core ASD symptoms. Based on strong preliminary evidence, this study aims to improve core ASD symptoms with folinic acid. Two biological mechanisms for response to the intervention are proposed and investigated in this study.

Folate is an essential B vitamin required for normal neurodevelopment. Folinic acid is a reduced form of folate that has been shown to improve both the metabolic and core symptoms associated with ASD in an open-label study and large case-series. This study will extend this preliminary evidence to demonstrate clinical efficacy of folinic acid in a double-blind placebo-controlled manner while also evaluating the biological mechanisms associated with the clinical response.

Preliminary evidence for the efficacy of folinic acid is two-fold: First, several independent studies have demonstrated that a folinic acid intervention improves ASD core symptoms in ASD patients diagnosed with cerebral folate deficiency - a metabolic disorder in which the primary pathway for the transport of folate across the blood-brain barrier is dysfunctional. The primary transport pathway for folate across the blood-brain barrier uses the folate receptor α (FRα) and energy dependent endocytosis. A secondary pathway, the reduced folate carrier (RFC), can transport reduced forms of folate, such as folinic acid, across the blood-brain barrier. In case-series of children with ASD and cerebral folate deficiency, folinic acid (0.5 to 2 mg/kg/day) improved communication, social interaction, attention, and stereotypical behavior in some (3-6) and completely ameliorated ASD symptoms in others (6, 7).

The major cause of cerebral folate deficiency is an autoantibody that binds to the FRα and interferes with its ability to bind and transport folate. Recently, Frye et al. found that (a) autoantibodies to the FRα were present in approximately 75% of children with ASD, and (b) an intervention with folinic acid (2mg/kg/day; max 50mg) in children with ASD and FRα autoantibodies resulted in significant improvements in parental ratings of receptive and expressive language, verbal communication, stereotypic behavior, and attention as compared to parental rating for children that did not undergo any intervention (wait group) over a similar time period. This proposal will extend these preliminary findings by documenting response to a folinic acid intervention in a double-blind placebo-controlled manner and test whether FRα autoantibody titers predict response to a folinic acid intervention. If FRα autoantibody titers are found to predict response to the intervention, such titers could provide a biomarker to identify a subset of children with ASD that may benefit from a folinic acid intervention and may even predict the development of ASD symptoms in high risk siblings during the presymptomatic period.

Second, the ratio of reduced-to-oxidized glutathione (GSH/GSSG) is an established measure of systemic redox status and oxidative stress that has been shown in three independent case-control studies to be significantly decreased in many ASD children. James et al. have shown in a 3 month open-label clinical trial that an intervention of folinic acid and methyl-B12 significantly improved GSH/GSSG and Vineland scores for expressive language, receptive language, and socialization in ASD children. Important unanswered questions are (a) whether this preliminary data can be confirmed in a larger double-blind placebo-controlled study, (b) whether redox status before the folinic acid intervention can predict response to intervention and (c) whether improved systemic redox status is associated with improvement in core ASD symptoms.

This study will assess whether a folinic acid intervention can improve both core symptoms of ASD (i.e., communication, socialization, stereotyped movements) and associated comorbid symptoms (i.e., attention) in a double-blind placebo controlled clinical trial. This study will address whether improvements in core ASD symptoms associated with the intervention are related to biomarkers of either (or both) biological mechanisms proposed to be influenced by the intervention (i.e., GSH/GSSG, FRα autoantibody titer). Thus, using these biomarkers, it may be possible that children with ASD who optimally respond to the folinic acid intervention can be readily identified early after diagnosis or even during the pre-symptomatic period.

This double blind, placebo-controlled (DBPC) study will evaluate the efficacy of Folinic Acid for the treatment of language impaired autism spectrum disorder patients aged 3-14 years. The study will consist of a single site trial with approximatley 48 entering the DBPC phase. Subjects will be male or female with current or prospective diagnosis of Autism Spectrum Disorder (ASD). Language Impairments will be defined by the CELF, or PLS when warranted.

Phase 1 will consist of approximately 57children aged 3-14 with a diagnosis of Autism Spectrum Disorder (as defined by the Autism Diagnostic Observation Schedule or the Autism Diagnostic Interview-Revised), until approximately 48 children with confirmed ASD are enrolled into a randomized control trial (RCT; Phase 2). Enrollment will continue as needed until approximately 43 complete Phase 2. Approximately 40 will enroll into phase 3.

Initial analyses will be undertaken to inspect data for errors, inconsistencies, and incomplete information. This will include examining the data with simple frequency tables and dot plots for univariate data and scatter plots and multi-way dot plots with bivariate and multivariate data. To summarize bivariate relationships among predictors and between predictors and outcomes, Spearman's rank correlation coefficient will be used. For reporting inferential statistics, regression coefficients along with the 95 percent confidence intervals will be used extensively to quantify degree of clinical importance.

The primary population will be the Intent-to-Treat (ITT) population and is defined as all subjects who have completed at least one post treatment primary outcome measure. A secondary analysis will be performed on the "as treated" population defined as those subjects who had at least 75% compliance of prescribed medications and have not significantly deviated from the protocol.

To determine whether the folinic acid intervention over a 12-week period improves core symptoms of autism spectrum disorder in Phase 2, the procedure Proc Mixed in SAS will be used to fit a mixed model analysis of covariance. For the multisite study, the full model with the response variable language assessment will include predictors such as: intervention, time, autoantibody, intervention by time interaction, autoantibody by intervention interaction, redox status, redox status by time interaction, and baseline covariates. However, for the single site study, the number of variables in the model will be limited due to the smaller sample size and separate models will be performed on subgroups to compare the effects of the treatment in various subgroups. The results from the mixed model will determine if the biomarkers of physiological abnormalities, both autoantibodies and redox status, predict intervention response. Similar analysis will be performed for the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria

* 1. Autism Spectrum Disorder (as defined by a gold standard measure for ASD diagnosis: the Autism Diagnostic Observation Schedule and/or Autism Diagnostic Interview-Revised). In an event where sufficient diagnostic information is lacking, and the PI believes that the clients meet all other inclusion criteria and a prospective diagnosis of an ASD is clinically warranted, and a formal diagnosis is scheduled to occur within a reasonable time frame from the date of study entry but before dispersing study drug/placebo, then the client may be considered as potentially eligible. Furthermore, a research-reliable rater must complete the diagnosis.
* 2. 3 years to 14 years of age
* 3. Language Impairment
* 4. Ability to maintain complementary, traditional, and/or behavioral interventions and to attempt to keep them constant during the study, when possible.
* 5. Unchanged complementary, traditional, and/or behavioral intervention for approximately 8 weeks prior to study entry, when possible.

Exclusion Criteria

* 1. Currently taking Antipsychotic medication
* 2. Vitamin or Element Supplementation that exceeds the IOM Tolerable Upper Intake Levels
* 3. Any moderate to severe positive response on that Aberrant Behavior Checklist Irritability subscale on questions: Injures self on purpose, is aggressive to other children or adults (verbally or physically), deliberately hurts himself/herself, and/or does physical violence to self.
* 4. Prematurity (<34 weeks gestation) as determined by medical history
* 5. Current uncontrolled gastroesophageal reflux or ongoing significant kidney or liver disease. The PI will determine whether any ongoing kidney or liver disease is significant.

  6. Drugs known to affect folate metabolism (e.g., methotrexate) and their derivatives.

  7. Profound sensory deficits (e.g. hearing and vision deficits) that could interfere with the interpretation of study results.

  8. Any major genetic defect, or mutation, that is known to be associated with disease or possibly related to disease that affects folate, methylation, and/or glutathione metabolism. Questions regarding eligibility concerning this criterion will be addressed with the lead site PI before enrollment into the trial.

  9. Documented current or active seizures, as defined by a clinical seizure or abnormal EEG within the past 6 months.

  10. Children with major single-gene abnormalities, such as Fragile X, Rett's Syndrome, etc., recognized chromosome syndromes, such as 15q11 microdeletion syndrome, or have been diagnosed with other well recognized syndromes, such as fetal alcohol syndrome. Children with copy number variants that represent known polymorphisms or benign changes will not be excluded. Questions regarding eligibility concerning this criterion should be addressed with the lead site PI before enrollment into the trial.

  11. Children diagnosed with congenital brain malformations, acquired brain insults, congenital or acquired microcephaly, or infection of the central nervous system.

  12. Children with major well-defined metabolic disease, such as mitochondrial disease, urea cycle disorders, succinic semialdehyde dehydrogenase deficiency, creatine deficiency syndromes, etc.

  13. Current therapies that could potentially interfere with interpretation of study results.

  14. Other conditions which, in the opinion of the study team, will place subjects at unacceptable risk or result in inability to interpret the study data.

  15. Unwillingness or inability to return for follow-up testing at specified interval.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, M.D./Ph.D., Principal Investigator — Director of Autism Research
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, Sailey A, Wynne R, Rose S, Melnyk S, Jill James S, Sequeira JM, Quadros EV. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Mol Psychiatry. 2018 Feb;23(2):247-256. doi: 10.1038/mp.2016.168. Epub 2016 Oct 18. PMID 27752075
- See also: If you have not signed up for the Arkansas Autism Alliance Registry, Sign up here!! — http://arkansasautismalliance.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study sponsor (UAMS) was unable to completely monitor the study or resolve outstanding queries. The study data cannot be fully validated by the sponsor. The study was placed on Full Clinical Hold by the FDA and terminated by the sponsor as a result of investigator non-compliance.
Period: Overall Study
Arm/Group | All Participants
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study sponsor (UAMS) was unable to completely monitor the study or resolve outstanding queries. The study data cannot be fully validated by the sponsor. The study was placed on Full Clinical Hold by the FDA and terminated by the sponsor as a result of investigator non-compliance.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Language Improvement
Description: Language (measured by the receptive and expressive CELF language index, and preschool language scale (PLS), as needed) will be the primary outcome for the study. Both preliminary studies have suggested that the folinic acid intervention will be associated with receptive and expressive language improvements.
Time Frame: (baseline and 12 weeks )
Population: as for baseline characteristics
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Improved Stereotyped Behavior and Improved Social Skills
Description: Stereotyped behavior (as measured by the OACIS (not at 6 weeks), ASQ, RBS-R, and ABC) and social skills (as measured by the Vineland (not at 6 weeks), ASQ, and SRS) will be the secondary outcomes.
Time Frame: (baseline, 6, and 12 weeks)
Population: No data because no patients were analyzed.
Arm/Group | Phase I | Phase II: 12 Week Folinic Acid or Placebo Intervention | Phase III: Open Label Extension of Folinic Acid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The study sponsor (UAMS) was unable to completely monitor the study or resolve outstanding queries. The study data cannot be fully validated by the sponsor. The study was placed on Full Clinical Hold by the FDA and terminated by the sponsor as a result of investigator non-compliance.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes